CLINICAL TRIAL: NCT06436443
Title: The Effect of SMS Counseling for Gestational Diabetes on Self-Efficacy and Knowledge Levels
Brief Title: SMS Counseling on Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Nurten Terkes, Principal Investigator, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MAKU GO 2020/193
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Gestational Diabetes
Keywords: Gestational diabetes mellitus,; Self-Efficacy,; SMS Counseling.
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Masking Description: Single (Participant) They did not know if they were in the control and intervention group at the time of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): In addition to routine physician check-ups, an SMS group was created for the individuals in the intervention group, and basic information messages for diabetes control were sent to this group at regular intervals. In addition, individuals asked questions via this group. At the end of the eight-week follow-up, the data collection forms were filled out again and the study was terminated.
  Interventions: Other: SMS Counseling
- Control Group (No Intervention): The same data collection forms were filled out at the first interview and eight weeks later by the pregnant women in the control group, and they continued to receive routine follow-ups.

INTERVENTIONS:
Other: SMS Counseling — In addition to routine physician check-ups, an SMS group was created for the individuals in the intervention group, and basic information messages for diabetes control were sent to this group at regular intervals. In addition, individuals asked questions via this group. At the end of the eight-week follow-up, the data collection forms were filled out again and the study was terminated.
  Arms: Intervention group

SUMMARY:
The use of technology-based education and counseling services in the self-management of gestational diabetes contributes to better control of blood sugar levels, motivation and increased self-efficacy in women. Therefore, this study was planned as interventional research to determine the effect of SMS counseling given to individuals with gestational diabetes on self-efficacy and knowledge levels. This study was conducted descriptively with 95 patients with gestational diabetes who were treated in the endocrine service of a university hospital between August 15, 2021 and April 24, 2022. Personal information form created by the researchers, The Self-Efficacy Scale in Gestational Diabetes, and Diabetes Knowledge Scale were used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with gestational diabetes,
* being in the 30th week of pregnancy,
* having a smartphone,
* volunteering to participate in the study,
* having no communication problems,
* having no psychiatric problems

Exclusion Criteria:

* being non-literate,
* having communication problems (hearing or sight),
* not volunteering to participate in the research

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women were taken.
Enrollment: 95 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-24 (Actual)

PRIMARY OUTCOMES:
Diabetes Knowledge Scale | 5 Minute
  This scale was first developed by Dunn et al.13 to measure diabetes knowledge. Afterward, it was developed by Carolan et al. to examine three effect domains: pregnant women's GDM knowledge, nutritional values, and GDM self-management principles. The scale consists of 18 questions. Cronbach's alpha value of the total scale was determined as 0.654.
The Self-Efficacy Scale in Gestational Diabetes | 5 minute
  This is a five-point Likert-type scale consisting of 23 items developed by Polat and Avdal in 2019 to evaluate the self-efficacy levels of individuals with gestational diabetes. It consists of four sub-dimensions: "diet-weight management"; "complication measures"; "compliance with nutrition education"; "medical therapy practices". As the total score on the scale increases, the level of self-efficacy increases, as well. Cronbach's alpha value of the total scale was determined as 0.654.

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All authors contributed to the interpretation, writing, and approval of the final manuscript.

REFERENCES:
- [Result] Hemmati Maslakpak M, Razmara S, Niazkhani Z. Effects of Face-to-Face and Telephone-Based Family-Oriented Education on Self-Care Behavior and Patient Outcomes in Type 2 Diabetes: A Randomized Controlled Trial. J Diabetes Res. 2017;2017:8404328. doi: 10.1155/2017/8404328. Epub 2017 Nov 22. PMID 29359166
- [Result] Guo Y, Zhou L, Sun B, Wang C, Zhang J. Application of online-offline integrated medical care management in patients with gestational diabetes. Ginekol Pol. 2021;92(10):720-725. doi: 10.5603/GP.a2021.0054. Epub 2021 Apr 29. PMID 33914304
- [Result] Miremberg H, Ben-Ari T, Betzer T, Raphaeli H, Gasnier R, Barda G, Bar J, Weiner E. The impact of a daily smartphone-based feedback system among women with gestational diabetes on compliance, glycemic control, satisfaction, and pregnancy outcome: a randomized controlled trial. Am J Obstet Gynecol. 2018 Apr;218(4):453.e1-453.e7. doi: 10.1016/j.ajog.2018.01.044. Epub 2018 Feb 7. PMID 29425836